CLINICAL TRIAL: NCT07138859
Title: Prospective, Multiceter, Randomized, Controlled Study on the Intraoperative Technical Errors of Robotic vs. Laparoscopic Radical Right Hemiclectomy (Superiority Design，ROBOGEON® 2501study)
Brief Title: The Intraoperative Technical Errors of Robotic vs. Laparoscopic Radical Right Hemiclectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Zhou Yanbing, Professor, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ROBOGEON 2501 study
Record Dates: First submitted 2025-07-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Carcinoma (CRC); Right Hemicolectomy
Keywords: Colorectal Carcinoma (CRC); right hemicolectomy; Robotic surgery; Errors; Intraoperative bleeding; Dangerous areas; Clinical outcome
MeSH Terms: conditions — Colorectal Neoplasms; Blood Loss, Surgical

STUDY DESIGN:
Masking Description: Video reviewers: 2 blind reviewers with at least 1000 hours of experience in reviewing surgical videos; The inter rater reliability between the two reviewers is over 85%; Complete human factors engineering training; A research committee composed of OC-HRA experts and consultant surgeons with OC-HRA experience conducted continuous inspections and supervision.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robot right hemicolectomy group (Experimental): Perform robot assisted radical right hemicolectomy (D3 lymph node dissection)
  Interventions: Device: Robot assisted radical right hemicolectomy (D3 lymph node dissection)
- Laparoscopic right hemicolectomy group (Active Comparator): Performing traditional laparoscopic radical right hemicolectomy (D3 lymph node dissection)
  Interventions: Device: Laparoscopic assisted radical right hemicolectomy (D3 lymph node dissection)

INTERVENTIONS:
Device: Robot assisted radical right hemicolectomy (D3 lymph node dissection) — RRH (Robotic Right Hemicolectomy) group: Experimental group: Performing robotic radical right hemicolectomy (D3 lymph node dissection)
  Arms: Robot right hemicolectomy group
Device: Laparoscopic assisted radical right hemicolectomy (D3 lymph node dissection) — LRH (Laparoscopic Right Hemicolectomy) group: control group: underwent laparoscopic radical right hemicolectomy (D3 lymph node dissection)
  Arms: Laparoscopic right hemicolectomy group

SUMMARY:
Experimental design: This study is a multicenter, prospective, randomized, controlled phase III clinical trial that identifies, classifies, defines, and quantitatively analyzes technical errors between robotic and laparoscopic radical right hemicolectomy (D3 lymph node dissection), identifies surgical risk areas, compares intraoperative performance, and patient short-term and long-term clinical outcomes.

This experimental design was based on a 1:1 effective target case ratio between the experimental group and the control group for enrollment. The experimental group underwent robotic radical right hemicolectomy (D3 lymph node dissection), while the control group underwent laparoscopic radical right hemicolectomy (D3 lymph node dissection). The unedited surgical videos of patients were analyzed, and relevant indicators and adverse events were recorded. Patients were followed up in the outpatient department after discharge until 3 years after surgery or until death or recurrence.

Sample size calculation: In this study, the calculation of sample size was based on pre experiments and hypotheses, and a goodness test was conducted by selecting the means of two independent samples. Referring to the results of the pilot study, based on a 1:1 random (random number table method) ratio, assuming a significance level of unilateral α=0.025, a test power of 1- β=80%, and a superiority margin of 20% in reducing the number of errors, and considering the maximum dropout rate of 0.1 in this clinical study, the total sample size for this study was determined to be 368 patients (184 in the RRC group and 184 in the LRC group).

Primary endpoint: incidence of technical errors during right hemicolectomy. Secondary endpoint: incidence of intraoperative complications; The incidence of complications within 30 days after surgery; Total surgical time, robot/laparoscope time; Estimate the amount of blood loss; Conversion to open surgery rate; Postoperative hospitalization time; Total number of lymph nodes cleared and positive rate of lymph nodes; Early postoperative recovery process (time of first defecation and defecation); 30 day readmission rate and unplanned reoperation rate after surgery; Postoperative nutritional status, inflammation, and immune response; 3-year disease-free survival rate DFS; 3-year overall survival rate (OS).

Inclusion criteria: 1) 18 years old<age<80 years old, regardless of gender; 2) The primary lesion of the colon was diagnosed as colon adenocarcinoma (well differentiated adenocarcinoma, moderately differentiated adenocarcinoma, poorly differentiated adenocarcinoma, mucinous adenocarcinoma) through endoscopic biopsy tissue pathology; 3) The preoperative clinical staging was cStage I-III (cT1-4a, N0/+, M0) (according to UICC/AJCC-8thTNM tumor staging); 4) The primary lesions of the colon are located in the cecum, ascending colon, hepatic flexure of the colon, and right half of the transverse colon. It is expected that right-sided colectomy and D3 lymph node dissection can achieve R0 surgical results (excluding multiple primary cancers); 5) Preoperative examination showed no distant metastasis, and the tumor did not directly invade adjacent organs; 6) Preoperative ECOG physical status score ≤ 2; 7) Preoperative ASA scores I-III; 8) Patient informed consent.

Exclusion criteria: 1) History of colon surgery (excluding ESD/EMR for colon cancer); 2) History of major abdominal surgery (excluding laparoscopic cholecystectomy and appendectomy); 3) Preoperative body temperature ≥ 38 ℃ or complicated with infectious diseases requiring systematic treatment; 4) Pregnant or lactating women; 5) Suffering from severe mental illness; 6) Multiple primary cancers; 7) History of other malignant diseases within 5 years; 8) Any neoadjuvant therapy such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc. has been implemented; 9) History of unstable angina or myocardial infarction within 6 months; 10) Heart, lung, liver, kidney dysfunction or history of cerebral infarction; 11) Simultaneous surgical treatment is required for other diseases; 12) Colorectal cancer complications (bleeding, perforation, obstruction) require emergency surgery.

DETAILED DESCRIPTION:
Right hemicolectomy and lymph node dissection scope: According to the Japanese Society for Colorectal Cancer Research (JSCCR) colon cancer treatment guidelines and the Chinese Society of Clinical Oncology (CSCO) colon cancer diagnosis and treatment guidelines, total mesorectal resection and D3 lymph node dissection are performed.

There are no requirements for digestive reconstruction methods, energy equipment, vascular ligation methods, gastrointestinal cutting and closure, digestive reconstruction instruments, or placement of abdominal drainage tubes.

Surgical task division

This study only records and analyzes the in vivo operation part (from Trocar insertion to CME release and vascular dissection), and does not require intestinal transverse and anastomosis methods, nor does it include statistical analysis. There are no specific requirements for the sequence of dissection and surgical operations. The main tasks can be divided into 5 parts:

1. Complete pneumoperitoneum - exposure of the surgical area.
2. Free posterior colon space (RRCS) and right colon:

   Find and open the Toldt gap, extend the gap until the dissociation of the right colon is completed. All operations in the RRCS area should belong to this recording section (right boundary: right colonic sulcus; left boundary: duodenal box; anterior: transverse mesentery; posterior: pre renal fascia).
3. Expose and ligate colon blood vessels or search for mesenteric blood vessels and open the vascular sheath, and clean lymph nodes:

   Expose and dissect the anterior part where the root of the colonic blood vessels merges into the SMV, ligate the colonic blood vessels, and perform root ligation on the right or main branch of the colonic blood vessels according to the tumor location. Expose the descending part of the duodenum and the head of the pancreas, dissect the SMV, and use the SMV as the inner boundary for lymph node dissection.
4. Open the gastrocolic ligament and search for the mesentery space:

   Open the root of the transverse colon mesentery and the gastrocolic ligament to fully free the transverse colon. During the process of drifting to the right, it is necessary to fully distinguish the gap between the transverse colon mesentery and the gastroduodenal mesentery.
5. Free transverse colon posterior space (TRCS) and anatomical Henle trunk:

Enter and maintain the TRCS until the branch dissection of the Henle trunk is completed. All operations involving the TRCS region (lateral boundary: descending segment of duodenum; medial boundary: superior mesenteric vein; head side: root of transverse mesentery; tail side boundary: horizontal part of duodenum; ventral boundary: dorsal side of transverse mesentery; dorsal side: anterior pancreatic fascia) and Henle trunk dissection should be included in this recording section.

Intraoperative bleeding grading Level 1: There is bleeding, but it does not affect the surgical operation and does not require any treatment; Level 2: Wound bleeding, unnamed vessel bleeding, clear surgical field of view, electrocoagulation, ultrasonic knife or compression hemostasis can all control bleeding without stopping the surgery; Grade III: Small vein bleeding, tear of liver, spleen, and pancreatic capsule, with no impact on hemodynamics. The surgical field of view is blurred, which affects the surgery, so it is necessary to stop the surgery to stop bleeding; Level 4: Bleeding from larger blood vessels and their branches, as well as the main blood vessels supplying the gastrointestinal tract, with hemodynamic fluctuations and ineffective compression hemostasis. Surgical hemostasis needs to be stopped, which can be controlled under the microscope and does not require conversion to open surgery; Grade 5: Bleeding from major blood vessels and their branches, as well as the main blood vessels supplying the gastrointestinal tract, with unstable hemodynamics, requiring a small amount of blood transfusion, uncontrollable under the microscope, and requiring conversion to open surgery for hemostasis. The patient's prognosis is good; Grade 6: Large abdominal blood vessels cause massive bleeding and have significant hemodynamic effects. A large amount of blood transfusion and vascular repair are required, which may lead to organ ischemia. The patient has a poor prognosis and may die.

Review of video footage. All unedited surgical videos are uploaded to the data platform of this study and handed over to two blind review expert reviewers with over 1000 hours of laparoscopic surgical video review experience in the surgical simulation laboratory of the Cuschieri Surgical Clinical Skills Training Center at the University of Dundee in the UK for identification, re coding, and analysis. Prior to the research, the reviewer completed 8 months of human factors engineering training under the guidance of clinical scientists at the University of Dundee's OC-HRA specialist (B.J.T.), which is a necessary prerequisite for proficient use of OC-HRA. Afterwards, reviewers and OC-HRA expert scientists independently analyzed ten videos of RRC and LRC. Ensure high inter rater reliability between the two reviewers. To ensure the accuracy of OC-HRA assessment video recordings, a research committee consisting of OC-HRA experts and experienced consultant surgeons conducted continuous inspections and supervision.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old<age<80 years old, regardless of gender;
2. The primary lesion of the colon was diagnosed as colon adenocarcinoma (well differentiated adenocarcinoma, moderately differentiated adenocarcinoma, poorly differentiated adenocarcinoma, mucinous adenocarcinoma) through endoscopic biopsy tissue pathology;
3. The preoperative clinical staging was cStage I-III (cT1-4a, N0/+, M0) (according to UICC/AJCC-8thTNM tumor staging);
4. The primary lesions of the colon are located in the cecum, ascending colon, hepatic flexure of the colon, and right half of the transverse colon. It is expected that right-sided colectomy and D3 lymph node dissection can achieve R0 surgical results (excluding multiple primary cancers);
5. Preoperative examination showed no distant metastasis, and the tumor did not directly invade adjacent organs;
6. Preoperative ECOG physical status score ≤ 2;
7. Preoperative ASA scores I-III;
8. Patient informed consent.

Exclusion Criteria:

1. History of colon surgery (excluding ESD/EMR for colon cancer);
2. History of major abdominal surgery (excluding laparoscopic cholecystectomy and appendectomy);
3. Preoperative body temperature ≥ 38 ℃ or complicated with infectious diseases requiring systematic treatment;
4. Pregnant or lactating women;
5. Suffering from severe mental illness;
6. Multiple primary cancers;
7. History of other malignant diseases within 5 years;
8. Any neoadjuvant therapy such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc. has been implemented;
9. History of unstable angina or myocardial infarction within 6 months;
10. Heart, lung, liver, kidney dysfunction or history of cerebral infarction;
11. Simultaneous surgical treatment is required for other diseases;
12. Colorectal cancer complications (bleeding, perforation, obstruction) require emergency surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Total number of technical errors during right hemicolectomy | Perioperative

SECONDARY OUTCOMES:
Incidence of intraoperative complications | Perioperative
Postoperative hospitalization time | Perioperative
Incidence of complications within 30 days after surgery | Within 30 days after surgery
3-year disease-free survival rate DFS | Within 3 years after surgery
Surgical time | Perioperative
estimated blood loss | Perioperative
conversion rate to open surgery | Perioperative
Early postoperative recovery process (time of first exhaust and defecation) | Perioperative
Postoperative nutritional status, inflammation, and immune response | Perioperative
Total number of lymph nodes cleared, positive rate of lymph nodes | Perioperative
readmission rate within 30 days after surgery | Within 30 days after surgery
unplanned reoperation rate within 30 days after surgery | Within 30 days after surgery
3-year overall survival rate OS | Within 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Shandong, Province, China

IPD SHARING:
Plan to Share IPD: Yes
The specific items of IPD planned for sharing are as follows:
  Demographic information: gender, age (years). Baseline characteristics: height, weight BMI、 Comorbidities (listed by ICD-10 code).
  Primary endpoint indicator:
  Number of intraoperative errors Secondary endpoint indicators;
  Intervention information:
  • Randomized grouping (experimental group/control group) Unshared data: directly identifiable personal information (name, address, phone number, complete date of birth, case number, original image files, etc.).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD First Sharing Start Date:
  The main research results are expected to be published in a peer-reviewed journal on March 1, 2028.
  End Date for IPD Sharing:
  The results will remain open for 5 years after publication, and sharing will be closed on March 1, 2033.
Access Criteria: Who: Qualified researchers with a scientifically valid proposal and documented approval from their local institutional review board (IRB) or ethics committee. Access is open to academic, non-profit, and regulatory entities; commercial organizations must provide a clear scientific rationale and sign the same data-use agreement (DUA).
  What:A fully de-identified dataset containing all efficacy, safety, and demographic variables specified in the protocol. Accompanying documents: protocol, statistical analysis plan (SAP), informed-consent form, data dictionary, blank and annotated case-report forms, and variable-coding manuals.
  How: Submit a brief research proposal plus IRB approval letter to the Data Sharing Committee via the secure portal. Data are downloaded as encrypted CSV/SAS transport files via a secure SFTP server; a remote virtual data enclave is also available for sensitive analyses. Data use is restricted to the approved project; any publication must cite the original trial.

REFERENCES:
- [Background] Tejedor P, Francis N, Jayne D, Hohenberger W, Khan J; on behalf the CME Project Working Group. Consensus statements on complete mesocolic excision for right-sided colon cancer-technical steps and training implications. Surg Endosc. 2022 Aug;36(8):5595-5601. doi: 10.1007/s00464-021-08395-0. Epub 2022 Jul 5. PMID 35790593
- [Background] Lu J, Xing J, Zang L, Zhang C, Xu L, Zhang G, He Z, Sun Y, Feng Y, Du X, Hu S, Chi P, Huang Y, Wang Z, Zhong M, Wu A, Zhu A, Li F, Xu J, Kang L, Suo J, Deng H, Ye Y, Ding K, Xu T, Zhang Y, Zhang Z, Zheng M, Su X, Xiao Y; RELARC study group. Extent of Lymphadenectomy for Surgical Management of Right-Sided Colon Cancer: The Randomized Phase III RELARC Trial. J Clin Oncol. 2024 Nov 20;42(33):3957-3966. doi: 10.1200/JCO.24.00393. Epub 2024 Aug 27. PMID 39190853
- [Background] Ahadi M, Sokolova A, Brown I, Chou A, Gill AJ. The 2019 World Health Organization Classification of appendiceal, colorectal and anal canal tumours: an update and critical assessment. Pathology. 2021 Jun;53(4):454-461. doi: 10.1016/j.pathol.2020.10.010. Epub 2021 Jan 16. PMID 33461799
- [Background] Gorard J, Boal M, Swamynathan V, Ghamrawi W, Francis N. The application of objective clinical human reliability analysis (OCHRA) in the assessment of basic robotic surgical skills. Surg Endosc. 2024 Jan;38(1):116-128. doi: 10.1007/s00464-023-10510-2. Epub 2023 Nov 6. PMID 37932602
- [Background] Tang B, Hanna GB, Joice P, Cuschieri A. Identification and categorization of technical errors by Observational Clinical Human Reliability Assessment (OCHRA) during laparoscopic cholecystectomy. Arch Surg. 2004 Nov;139(11):1215-20. doi: 10.1001/archsurg.139.11.1215. PMID 15545569
- [Background] Foster JD, Miskovic D, Allison AS, Conti JA, Ockrim J, Cooper EJ, Hanna GB, Francis NK. Application of objective clinical human reliability analysis (OCHRA) in assessment of technical performance in laparoscopic rectal cancer surgery. Tech Coloproctol. 2016 Jun;20(6):361-367. doi: 10.1007/s10151-016-1444-4. Epub 2016 May 6. PMID 27154295
- [Background] Dyreborg J, Lipscomb HJ, Nielsen K, Torner M, Rasmussen K, Frydendall KB, Bay H, Gensby U, Bengtsen E, Guldenmund F, Kines P. Safety interventions for the prevention of accidents at work: A systematic review. Campbell Syst Rev. 2022 Jun 1;18(2):e1234. doi: 10.1002/cl2.1234. eCollection 2022 Jun. PMID 36911341
- [Background] Miskovic D, Ni M, Wyles SM, Parvaiz A, Hanna GB. Observational clinical human reliability analysis (OCHRA) for competency assessment in laparoscopic colorectal surgery at the specialist level. Surg Endosc. 2012 Mar;26(3):796-803. doi: 10.1007/s00464-011-1955-z. Epub 2011 Nov 1. PMID 22042584
- [Background] Jia Z, Cao S, Wang D, Tang C, Tan X, Liu S, Liu X, Li Z, Tian Y, Niu Z, Tang B, Zhou Y. Identification and Categorization of Technical Errors and Hazard Zones of Robotic Versus Laparoscopic Total Gastrectomy for Gastric Cancer: A Single-center Prospective Randomized Controlled Study. Ann Surg. 2025 Jul 1;282(1):37-45. doi: 10.1097/SLA.0000000000006585. Epub 2024 Nov 8. PMID 39513271
- [Background] Kitz J, Fokas E, Beissbarth T, Strobel P, Wittekind C, Hartmann A, Ruschoff J, Papadopoulos T, Rosler E, Ortloff-Kittredge P, Kania U, Schlitt H, Link KH, Bechstein W, Raab HR, Staib L, Germer CT, Liersch T, Sauer R, Rodel C, Ghadimi M, Hohenberger W; German Rectal Cancer Study Group. Association of Plane of Total Mesorectal Excision With Prognosis of Rectal Cancer: Secondary Analysis of the CAO/ARO/AIO-04 Phase 3 Randomized Clinical Trial. JAMA Surg. 2018 Aug 1;153(8):e181607. doi: 10.1001/jamasurg.2018.1607. Epub 2018 Aug 15. PMID 29874375
- [Background] Curtis NJ, Dennison G, Brown CSB, Hewett PJ, Hanna GB, Stevenson ARL, Francis NK. Clinical Evaluation of Intraoperative Near Misses in Laparoscopic Rectal Cancer Surgery. Ann Surg. 2021 Apr 1;273(4):778-784. doi: 10.1097/SLA.0000000000003452. PMID 31274657
- [Background] Zhang Y, Feng H, Wang S, Gu Y, Shi Y, Song Z, Deng Y, Ji X, Cheng X, Zhang T, Zhao R. Short- and long-term outcomes of robotic- versus laparoscopic-assisted right hemicolectomy: A propensity score-matched retrospective cohort study. Int J Surg. 2022 Sep;105:106855. doi: 10.1016/j.ijsu.2022.106855. Epub 2022 Aug 24. PMID 36030038
- [Background] Clarke EM, Rahme J, Larach T, Rajkomar A, Jain A, Hiscock R, Warrier S, Smart P. Robotic versus laparoscopic right hemicolectomy: a retrospective cohort study of the Binational Colorectal Cancer Database. J Robot Surg. 2022 Aug;16(4):927-933. doi: 10.1007/s11701-021-01319-z. Epub 2021 Oct 28. PMID 34709537
- [Background] de'Angelis N, Schena CA, Espin-Basany E, Piccoli M, Alfieri S, Aisoni F, Coccolini F, Frontali A, Kraft M, Lakkis Z, Le Roy B, Luzzi AP, Milone M, Pattacini GC, Pellino G, Petri R, Piozzi GN, Quero G, Ris F, Winter DC, Khan J; MERCY Study Collaborating Group Members. Robotic versus laparoscopic right colectomy for nonmetastatic pT4 colon cancer: A European multicentre propensity score-matched analysis. Colorectal Dis. 2024 Aug;26(8):1569-1583. doi: 10.1111/codi.17089. Epub 2024 Jul 8. PMID 38978153
- [Background] Formisano G, Misitano P, Giuliani G, Calamati G, Salvischiani L, Bianchi PP. Laparoscopic versus robotic right colectomy: technique and outcomes. Updates Surg. 2016 Mar;68(1):63-9. doi: 10.1007/s13304-016-0353-4. Epub 2016 Mar 18. PMID 26992927
- [Background] Zelhart M, Kaiser AM. Robotic versus laparoscopic versus open colorectal surgery: towards defining criteria to the right choice. Surg Endosc. 2018 Jan;32(1):24-38. doi: 10.1007/s00464-017-5796-2. Epub 2017 Aug 15. PMID 28812154
- [Background] Franklin A, Patterson A, Taylor J, Avery M, Pullatt R. Laparoscopic Right Hemicolectomy in a Morbidly Obese Patient Using a Medial Approach with an Intracorporeal Anastomosis. Am Surg. 2015 Aug;81(8):301-2. No abstract available. PMID 26215227
- [Background] Matsuda T, Yamashita K, Hasegawa H, Utsumi M, Kakeji Y. Current status and trend of laparoscopic right hemicolectomy for colon cancer. Ann Gastroenterol Surg. 2020 Jul 18;4(5):521-527. doi: 10.1002/ags3.12373. eCollection 2020 Sep. PMID 33005847
- [Background] Lee CZ, Kao LT, Lin HC, Wei PL. Comparison of clinical outcome between laparoscopic and open right hemicolectomy: a nationwide study. World J Surg Oncol. 2015 Aug 15;13:250. doi: 10.1186/s12957-015-0666-7. PMID 26271770
- [Background] Zhao LY, Chi P, Ding WX, Huang SR, Zhang SF, Pan K, Hu YF, Liu H, Li GX. Laparoscopic vs open extended right hemicolectomy for colon cancer. World J Gastroenterol. 2014 Jun 28;20(24):7926-32. doi: 10.3748/wjg.v20.i24.7926. PMID 24976728
- [Background] Kahokehr A, Sammour T, Zargar-Shoshtari K, Srinivasa S, Hill AG. Recovery after open and laparoscopic right hemicolectomy: a comparison. J Surg Res. 2010 Jul;162(1):11-6. doi: 10.1016/j.jss.2010.02.008. Epub 2010 Mar 9. PMID 20452623
- [Background] Kim HS, Noh GT, Chung SS, Lee RA. Long-term oncological outcomes of robotic versus laparoscopic approaches for right colon cancer: a systematic review and meta-analysis. Tech Coloproctol. 2023 Dec;27(12):1183-1189. doi: 10.1007/s10151-023-02857-4. Epub 2023 Oct 3. PMID 37783821
- [Background] Mitchell BG, Mandava N. Hemicolectomy. 2023 Jun 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK555924/ PMID 32310384
- [Background] Yuval JB, Thompson HM, Verheij FS, Fiasconaro M, Patil S, Widmar M, Wei IH, Pappou EP, Smith JJ, Nash GM, Weiser MR, Paty PB, Garcia-Aguilar J. Comparison of Robotic, Laparoscopic, and Open Resections of Nonmetastatic Colon Cancer. Dis Colon Rectum. 2023 Oct 1;66(10):1347-1358. doi: 10.1097/DCR.0000000000002637. Epub 2022 Dec 16. PMID 36649145
- [Background] Lygre KB, Eide GE, Forsmo HM, Dicko A, Storli KE, Pfeffer F. Complications after open and laparoscopic right-sided colectomy with central lymphadenectomy for colon cancer: randomized controlled trial. BJS Open. 2023 Jul 10;7(4):zrad074. doi: 10.1093/bjsopen/zrad074. PMID 37643373
- [Background] Lovay K, Barla J, Vasko J, Lendel A, Rakos M. Laparoscopic versus open elective right hemicolectomy with curative intent for colon adenocarcinoma. Rozhl Chir. 2022 Winter;100(12):584-591. doi: 10.33699/PIS.2021.100.12.584-591. PMID 35042343
- [Background] Vogel JD, Felder SI, Bhama AR, Hawkins AT, Langenfeld SJ, Shaffer VO, Thorsen AJ, Weiser MR, Chang GJ, Lightner AL, Feingold DL, Paquette IM. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Management of Colon Cancer. Dis Colon Rectum. 2022 Feb 1;65(2):148-177. doi: 10.1097/DCR.0000000000002323. No abstract available. PMID 34775402
- [Background] Parkin DM, Muir CS. Cancer Incidence in Five Continents. Comparability and quality of data. IARC Sci Publ. 1992;(120):45-173. No abstract available. PMID 1284606
- [Background] Menon G, Cagir B. Colon Cancer. 2025 Feb 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470380/ PMID 29262132